CLINICAL TRIAL: NCT02343107
Title: E-coaching for Patients With Abdominal Obesity and Type 2 Diabetes : the A.N.O.D.E. Study
Brief Title: E-coaching for Type 2 Diabetes
Acronym: ANODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K120901
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2015-07

CONDITIONS: Abdominal Obesity; Type 2 Diabetes
Keywords: Obesity; Type 2 diabetes; Metabolic syndrome; e-coaching; Telehealth
MeSH Terms: conditions — Obesity, Abdominal; Diabetes Mellitus, Type 2; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subgroup of subjects who benefit of the e-coaching
  Interventions: Behavioral: e-coaching
- 2 (No Intervention): Subgroup of subjects who are asked to follow the conventional nutritional recommendations of the treatment of abdominal obesity and diabetes

INTERVENTIONS:
Behavioral: e-coaching — connexion to a website and interaction with an automatizes system which delivers tailored recommendations over a 4 month period.
  Arms: 1

SUMMARY:
Abdominal obesity and its metabolic consequences, particularly type 2 diabetes, require personalized nutritional monitoring. Today, it is not always possible to provide patients with appropriate care to both, the diet plan, physical activity, stress and sleep management. Emerging data have shown the effectiveness of remote support (e- coaching), in order to increase the level of physical activity and reducing calorie intake which causes weight loss similar to that obtained during a face to face consultation. Compared to a food survey conducted by a dietician, the dietary survey MXS computer software showed similar results on the collection of nutritional data. Furthermore, users preferred this method of remote collection compared to direct interview. The investigators recently developed a tool for e-coaching combining this computerized dietary survey and education and support modules on diet and physical activity (MXS- health program) for the patients. The aim of the investigators' study is to compare efficacy of this new software vs usual care.

DETAILED DESCRIPTION:
Description of nutritional intervention in both groups:

Both groups make the same visits, answer the same questionnaire and dietary surveys. Only nutrition and physical activity recommendations differ depending on whether the patient is randomized to the intervention group or the control group.

* Intervention group: e-coaching: patients benefit from the MXS-health support program including self-monitoring modules, generation of adequate nutritional recipes, education and support for physical activity. They receive an access code and personal password during the randomization visit
* Control group: usual recommendations: Control subjects will simply follow the usual nutritional recommendations provided during the monitoring of their diabetes. They will be informed of the possibility to benefit from the e-coaching program at the end of the study.

Research hypotheses

Assumptions related to this research are :

* The MXS -health e-coaching program improves adherence to nutritional recommendations in patients with abdominal obesity and type 2 diabetes.
* Adhesion to the e-coaching program can be predicted by simple criteria based on the characteristics of the patient and a self-administered questionnaire including socio-professional characteristics and the level of food impulsivity.

Main objective To show that within four months, the e-coaching improves eating habits. The primary endpoint is the comparison of the changes between the first (D-20 D-2) and the second survey (D100 to D118) of dietary score (International Diet Quality Index) between both groups (e-coaching versus usual nutritional recommendations).

Secondary objectives

* To show that the e-coaching provides in four months, an increase in both duration and abilities for physical activity,
* To identify predictors of the effectiveness and adherence to the e-coaching program which take into account the average number of weekly connections and the percentage of tasks required by the software (watch a video, fill a questionnaire ...) performed by the included patients,
* To evaluate the effectiveness of e-coaching on glycaemic control (HbA1c) and the cardiometabolic risk profile (lipid parameters, blood pressure, waist circumference, weight, hs-CRP, transaminases, adiponectin),
* To evaluate the effectiveness of e-coaching on physical fitness (VO2 max calculated during a graded exercise test) and the amount of physical activity performed (IPAQ questionnaires).

ELIGIBILITY:
Inclusion criteria :

* Subject, male or female, aged 18-75 years (inclusive) who agrees to participate in the study and who gave verbal consent
* Abdominal obesity defined by waist circumference ≥ 102 cm for men and ≥ 88 cm for women
* Diabetic subject with HbA1C between 5,6% and 8,5% in the month before selection (using venous or capillary blood samples)
* Subject have already received a standard nutrition education for the treatment of diabetes
* Initial Food survey showing an estimated average calorie intake between 1200 and 4000 calories
* Anti-diabetic treatments, antihypertensive or lipid-lowering therapy stable for at least 3 months (at the initial blood test)
* Subject of a weight and a stable diet, not restrictive in the past 3 months (weight change ≤ 4 kg peak to peak)
* Affiliated to the social security system or having a similar regime
* Access to Internet and usual use, possession of an email address
* Understanding and reading French

Exclusion criteria :

* Excessive alcohol consumption (> 30 g / day on average)
* Symptomatic cardiovascular disease (myocardial infarction, angina pectoris, surgical or endovascular intervention, stroke older than 6 months, symptomatic lower limb arteritis)
* Subject receiving general or local treatment that may interfere with the assessment of the primary endpoint
* Situation requiring rapid equilibration of diabetes
* Subject with any severe or acute illness which may influence the results of the study or to life-threatening
* Subject in a situation which, in the opinion of the investigator, would interfere with the optimal participation in the study or be a particular risk for the patient
* Patient who underwent obesity surgery to the exclusion of a gastric band, loosened or removed for more than a year
* For female subjects: pregnancy or lactation, or subject may become pregnant during the study
* For female subjects: subject may change hormone treatment under study (contraceptive or hormone replacement)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
dietary score (International Diet Quality Index) | 4 months
  Comparison of the changes between the first (D-20 D-2) and the second survey (D100 to D118) of dietary score (International Diet Quality Index) between both groups (e-coaching versus usual nutritional recommendations).

SECONDARY OUTCOMES:
Physical skills measured by VO2max | 4 months
  Variation between D0 (± 8d)) and D120-D140 of Physical skills measured by VO2max
Physical activity (self-administered questionnaire IPAQ) | 4 months
  Variation between D0 (± 8d)) and D120-D140 of Physical activity (self-administered questionnaire IPAQ)
Weight | 4 months
  Variation between D0 (± 8d)) and D120-D140 of Weight
waist circumference | 4 months
  Variation between D0 (± 8d)) and D120-D140 of waist circumference
Biological parameters: Biological parameters: HbA1c, triglycerides, HDL-C, LDL-C, AST, ALT, uric acid, hs-CRP, adiponectin | 4 months
  Variation between D0 (± 8d)) and D120-D140 of Biological parameters: HbA1c, triglycerides, HDL-C, LDL-C, AST, ALT, uric acid, hs-CRP, adiponectin
Blood pressure | 4 months
  Variation between D0 (± 8d)) and D120-D140 of Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Boris Hansel, MD, PhD, Principal Investigator — Asistance Publique - Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpetrière, Paris, France

REFERENCES:
- [Result] Hansel B, Giral P, Gambotti L, Lafourcade A, Peres G, Filipecki C, Kadouch D, Hartemann A, Oppert JM, Bruckert E, Marre M, Bruneel A, Duchene E, Roussel R. A Fully Automated Web-Based Program Improves Lifestyle Habits and HbA1c in Patients With Type 2 Diabetes and Abdominal Obesity: Randomized Trial of Patient E-Coaching Nutritional Support (The ANODE Study). J Med Internet Res. 2017 Nov 8;19(11):e360. doi: 10.2196/jmir.7947. PMID 29117929